CLINICAL TRIAL: NCT06629870
Title: Evaluation of the Effect of Hypnotherapy, Virtual Reality and Mindfulness Applications on Dental Anxiety During Restorative Dental Treatment
Brief Title: Dental Anxiety During Restorative Dental Treatment
Acronym: DADRDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Fatih Alkan, Research assistant dentist, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATAUNIRESTORATIVE1
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Hypnotherapy; Virtual Reality; Mindfulness
Keywords: Dental anxiety, hypnotherapy, virtual reality glasses application, mindfulness-based meditation practice
MeSH Terms: interventions — Control Groups; Hypnosis; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator)
  Interventions: Other: control group
- hypnotherapy (Active Comparator)
  Interventions: Other: hypnotherapy
- virtual reality (Active Comparator)
  Interventions: Device: virtual reality
- mindfulness-based meditation (Active Comparator)
  Interventions: Other: mindfulness

INTERVENTIONS:
Device: virtual reality — patients who received distraction using virtual reality glasses
  Arms: virtual reality
Other: control group — no any anxiety-reducing application
  Arms: Control
Other: hypnotherapy — patients receiving hypnotherapy
  Arms: hypnotherapy
Other: mindfulness — patients who underwent mindfulness-based meditation
  Arms: mindfulness-based meditation

SUMMARY:
Anxiety refers to behavioural disorders associated with excessive fear and anxiety. Dental anxiety refers to excessive fear and anxiety at the thought of going to the dentist. This may cause patients to avoid dental treatments and may adversely affect oral health.

This study aims to evaluate the effects of hypnotherapy, virtual reality distraction and mindfulness-based meditation practices on dental anxiety during restorative dental treatment.

ELIGIBILITY:
Inclusion Criteria:

* A modified dental anxiety score of 20 and above
* A dental fear scale score of 59 and above
* D2 level caries according to radiographic caries classification system,
* Systemically healthy patients

Exclusion Criteria:

* Balance disorders such as nystagmus and vertigo,
* Pregnant woman
* Claustrophobia
* Physical or mental disability
* Not knowing how to read and write
* Psychological disturbance
* Taking antidepressants or anxiolytics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-26 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Modified Dental Anxiety Scale | 5 minutes before procedure and 5 minutes after procedure
  The Modified Dental Anxiety Scale (MDAS) consists of 5 questions each with a 5 category rating scale, ranging from 'not anxious' to 'extremely anxious'.

SECONDARY OUTCOMES:
Dental Fear Survey | 5 minutes before procedure and 5 minutes after procedure
  The items in this questionnaire refer to various situations, feelings, and reactions related to dental work
The Visual Analogue Scale | 5 minutes after procedure
  The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Faculty of Dentistry, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Joda T, Gallucci GO, Wismeijer D, Zitzmann NU. Augmented and virtual reality in dental medicine: A systematic review. Comput Biol Med. 2019 May;108:93-100. doi: 10.1016/j.compbiomed.2019.03.012. Epub 2019 Mar 15. PMID 31003184
- [Result] Prado IM, Carcavalli L, Abreu LG, Serra-Negra JM, Paiva SM, Martins CC. Use of distraction techniques for the management of anxiety and fear in paediatric dental practice: A systematic review of randomized controlled trials. Int J Paediatr Dent. 2019 Sep;29(5):650-668. doi: 10.1111/ipd.12499. Epub 2019 Apr 25. PMID 30908775